CLINICAL TRIAL: NCT03774186
Title: Pregnancy Intervention With a Closed-Loop System (PICLS) Study
Acronym: PICLS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: Juvenile Diabetes Research Foundation (Other); Ohio State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 18-1798
Record Dates: First submitted 2018-12-05; First posted 2018-12-12 (Actual); Results first posted 2023-11-28 (Actual); Last update posted 2023-11-28 (Actual); Status verified 2023-11

CONDITIONS: Type 1 Diabetes Mellitus; Pregnancy in Diabetes
Keywords: type 1 diabetes mellitus; pregnancy; hybrid closed-loop therapy; artificial pancreas therapy; sensor-augmented pump therapy
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Pregnancy in Diabetics

STUDY DESIGN:
Intervention Model Description: Randomized clinical trial
Who Masked: Outcomes Assessor
Masking Description: Biostatistician is blinded to intervention assignment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Sensor-augmented pump therapy (SAPT) (Active Comparator): Pregnant women with T1D with use an insulin pump and a continuous glucose monitor but there will be no automated insulin adjustments made by the system.
  Interventions: Device: Sensor-augmented pump therapy
- Hybrid closed-loop therapy (HCL) (Experimental): Pregnant women with T1D with use an insulin pump and a continuous glucose monitor with automated insulin adjustments made by the system, but continued meal boluses from the women.
  Interventions: Device: Hybrid closed-loop therapy

INTERVENTIONS:
Device: Hybrid closed-loop therapy — Hybrid closed-loop therapy with a proportional integral derivative (PID) algorithm
  Other Names: artificial pancreas therapy
  Arms: Hybrid closed-loop therapy (HCL)
Device: Sensor-augmented pump therapy — Insulin pump + non-communicating CGM
  Other Names: SAPT
  Arms: Sensor-augmented pump therapy (SAPT)

SUMMARY:
In pregnancies associated with diabetes, lowering glucose to the recommended targets to prevent adverse health outcomes often leads to significant hypoglycemia. Hybrid closed-loop (HCL) therapy, automated insulin delivery using an insulin pump getting feedback from a continuous glucose monitor (CGM), may improve outcomes. This exploratory, novel pilot feasibility randomized clinical trial will evaluate pregnant women with type 1 diabetes (T1D) on HCL therapy or Sensor-Augmented Pump Therapy (SAPT, non-communicating pump and CGM) from the 2nd trimester, throughout pregnancy, and 4-6 weeks post-partum. Comparisons will be made on safety (Specific Aim [SA] 1), indices of glycemic variability and fear of hypoglycemia (SA 2), and quality of life and device satisfaction (SA 3) between groups. Exploratory SA 4 will compare maternal and fetal outcomes between groups. Safety data will include episodes of severe hypoglycemia requiring 3rd party assistance, diabetic ketoacidosis, and skin reactions. Glycemic control will be measured by CGM time spent in glucose ranges (<63, 63-140, >140 mg/dL) and other measures of glycemic variability. Subjects will fill out surveys (Fear of Hypoglycemia, a quality of life survey, and 2 questionnaires about device satisfaction) at baseline, throughout gestation, and early post-partum. Data on maternal and fetal outcomes will be collected. Findings will reveal the safety profile and glucose control with a novel therapy for pregnant women with type 1 diabetes.

DETAILED DESCRIPTION:
This is a two-center, prospective, 'open-label', single-blind, investigator-initiated randomized controlled pilot study evaluating hybrid closed-loop (HCL) insulin delivery among pregnant women with T1D compared with sensor-augmented pump therapy (SAPT) throughout most of gestation and the first 6 weeks of the post-partum period at the Barbara Davis Center for Diabetes and Ohio State University.

Up to 37 women will be enrolled at ≤11 weeks gestation, sign informed consent, and begin a run-in phase. At baseline, the investigators will obtain data about demographics, health history, pregnancy history, and medication use. The investigators will conduct a physical exam, download diabetes devices already in use by subjects, obtain blood and urine tests, and administer validated questionnaires (Hypoglycemia Fear Survey, MOS Short-Form 36 [SF-26], INSPIRE Questionnaire, Insulin Delivery Satisfaction Survey [IDSS], and Glucose Monitoring Satisfaction Survey [GMSS]). During run-in, women will wear a CGM, fill out log sheets (glucose levels, insulin doses, carbohydrate intake, exercise), upload the CGM, and be in contact with research staff. Eligible subjects will then be trained on study devices for SAPT therapy. At the start of the 2nd trimester, women will be randomized to SAPT or HCL therapy.

During pregnancy, women will be seen at each institution monthly for vital signs, HbA1c measurements, device downloads, pump adjustments, medication use, reporting of adverse events and device-related deficiencies, and once a trimester the investigators will additionally obtain serum and urine measurements, specimens for the repository of biological specimens, and ask subjects to fill out questionnaires (Hypoglycemia Fear Survey, SF-35, IDSS, GMSS). Weekly remote contact will be obtained for pump adjustments and reporting of adverse events and device-related deficiencies. Women on HCL therapy will use SAPT during labor and delivery until 3-7 days post-partum, when a study clinician will put them back into auto mode (HCL therapy), if it is safe to do so. The final study visit will take place 4-6 weeks post-partum where the physical exam will be done, HbA1c obtained, device downloads obtained, and final questionnaires submitted (as above plus a post-partum survey). Medical records of the labor and delivery admission will be obtained.

ELIGIBILITY:
Inclusion Criteria:

* women with T1D,
* pregnant within the first 11 weeks of gestation,
* 18 years of age or older,
* diabetes duration >1 year,
* using MDI (multiple daily injections) or CSII (continuous subcutaneous insulin infusion) therapy,
* willingness to routinely check at least 3-7 blood glucose measurements per day,
* ability and willingness to receive routine and specialty obstetric care throughout the course of the study,
* ability and willingness to adhere to the protocol including scheduled study visits for the duration of the pregnancy and early post-partum period,
* A1C 5.5 - 9%,
* willing to participate in the run-in phase and full study (if eligible), and
* able to speak, read, and write English

Exclusion Criteria:

* women with T2D, gestational diabetes, or other type of diabetes (e.g., MODY), - -
* pregnancy beyond gestational week 11 or higher,
* age <18 years,
* T1D duration <1 year,
* screening A1C <5.5% or >9%,
* use of basal insulin alone,
* use of bolus insulin alone,
* extensive skin changes/diseases that inhibit wearing an infusion set, insulin pod, or sensor on normal skin,
* known severe allergic reaction to device adhesives within the last 3 months,
* unwillingness to use an insulin pump with tubing,
* unwillingness to be randomized to study group,
* unwillingness to switch from MDI to CSII and CGM (continuous glucose monitor) use (if applicable),
* unwillingness to switch from MDI or to change from current insulin pump to HCL system (if applicable),
* severe hypoglycemic episode requiring the assistance of a 3rd party within the last 6 months,
* non-compliance with run-in phase,
* inadequate access to a phone and computer (for downloading devices and web-based communications),
* intention to move out of state within the next year, and
* any other condition determined by the PI which could make the subject unsuitable for the trial or impairs the validity of the informed consent

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2019-03-21 (Actual); Primary Completion 2022-03-08 (Actual); Study Completion 2022-03-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sarit Polsky, MD, MPH, Principal Investigator — Regents of the University of Colorado
Locations (2):
- United States (2):
  - University of Colorado, Aurora, Colorado
  - Ohio State University Wexner Medical Center, Columbus, Ohio

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Sensor-augmented Pump Therapy (SAPT) | Hybrid Closed-loop Therapy (HCL)
Started | 12 | 12
Completed | 12 | 11
Not Completed | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sensor-augmented Pump Therapy (SAPT) | Hybrid Closed-loop Therapy (HCL) | Total
Number analyzed (Participants) | 12 | 12 | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.7 (3.5) | 31.5 (4.9) | 31.1 (4.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 12 | 24
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: Data not available for 3 participants
  Participants
    Non Hispanic White: number analyzed (Participants) | 10 | 11 | 21
    Non Hispanic White | 10 | 11 | 21
Education [Count of Participants; unit: Participants] — Population: Data missing for 1 in SAPT Group
  Participants
    number analyzed (Participants) | 11 | 12 | 23
    High School/General Education Development | 0 | 1 | 1
    Some College | 3 | 0 | 3
    Associate's Degree | 0 | 0 | 0
    Bachelor's Degree | 5 | 6 | 11
    Master's Degree | 2 | 5 | 7
    Doctorate | 1 | 0 | 1
Insurance Type [Count of Participants; unit: Participants]
  Medicaid | 0 | 1 | 1
  Government | 1 | 1 | 2
  Commercial | 8 | 5 | 13
  Other | 3 | 5 | 8
Multiparity [Count of Participants; unit: Participants] | 7 | 8 | 15
Tobacco Use [Count of Participants; unit: Participants] — Population: Missing data for 1 in SAPT Group
  Participants
    number analyzed (Participants) | 11 | 12 | 23
    Former | 3 | 1 | 4
    Never | 8 | 11 | 19
Insulin Pump Use Prior to Pregnancy [Count of Participants; unit: Participants] | 11 | 12 | 23
CGM Use Prior to Pregnancy [Count of Participants; unit: Participants] | 11 | 12 | 23

OUTCOME MEASURES:

1. Primary Outcome: Number of Episodes of Severe Hypoglycemia
Description: Safety of HCL therapy compared to SAPT in women with T1D throughout gestation and the early post-partum period assessed through the number of episodes of severe hypoglycemia requiring 3rd party assistance
Time Frame: through study completion, an average of 9 months
Measure: Number; unit: Number of Episodes
Arm/Group | Sensor-augmented Pump Therapy (SAPT) | Hybrid Closed-loop Therapy (HCL)
Number analyzed (Participants) | 12 | 11
Number of Episodes | 0 | 0

2. Primary Outcome: Time Spent With Glucose <54 mg/dL
Description: Safety of HCL therapy compared to SAPT in women with T1D throughout gestation and the early post-partum period assessed through continuous glucose monitor time spent with glucose <54 mg/dL
Time Frame: Through study completion, an average of 9 months
Measure: Mean (Standard Error); unit: percentage of time spent in range
Arm/Group | Sensor-augmented Pump Therapy (SAPT) | Hybrid Closed-loop Therapy (HCL)
Number analyzed (Participants) | 12 | 11
percentage of time spent in range
  Time spent with glucose <54 mg/dL (1st Trimester) | 3.98 (0.668) | 4.04 (0.683)
  Time spent with glucose <54 mg/dL (2nd Trimester) | 2.84 (0.668) | 1.68 (0.683)
  Time spent with glucose <54 mg/dL (3rd Trimester) | 2.01 (0.668) | 1.23 (0.683)
  Time spent with glucose <54 mg/dL (Postpartum) | 2.66 (0.679) | 1.16 (0.683)

3. Primary Outcome: Indices of Glucose Control: Time Spent in Glucose Ranges by Continuous Glucose Monitoring
Description: Indices of glucose control are time spent in the glucose target ranges <54 mg/dL and <63 mg/dL (hypoglycemia), 63-140 mg/dL (time in range), and >140 mg/dL and >180 mg/dL (hyperglycemia) of HCL compared to SAPT in women with T1D throughout gestation and the first 4-6 weeks post-partum
Time Frame: Through study completion, an average of 9 months
Measure: Mean (Standard Error); unit: percentage of time spent in range
Arm/Group | Sensor-augmented Pump Therapy (SAPT) | Hybrid Closed-loop Therapy (HCL)
Number analyzed (Participants) | 12 | 11
percentage of time spent in range
  Time spent <54 mg/ dL (1st Trimester) | 3.98 (0.668) | 4.04 (0.683)
  Time spent <54 mg/ dL (2nd Trimester) | 2.84 (0.668) | 1.68 (0.683)
  Time spent <54 mg/ dL (3rd Trimester) | 2.01 (0.668) | 1.23 (0.683)
  Time spent <54 mg/ dL (Postpartum) | 2.66 (0.679) | 1.16 (0.683)
  Time spent <63 mg/ dL (1st trimester) | 8.07 (1.15) | 7.46 (1.18)
  Time spent <63 mg/ dL (2nd trimester) | 6.26 (1.15) | 3.52 (1.18)
  Time spent <63 mg/ dL (3rd trimester) | 5.05 (1.15) | 2.81 (1.18)
  Time spent <63 mg/ dL (Postpartum) | 5.60 (1.17) | 2.58 (1.18)
  Time spent 63-140 mg/ dL (1st Trimester) | 62.2 (2.95) | 61.7 (3.02)
  Time spent 63-140 mg/ dL (2nd Trimester) | 60.6 (2.95) | 57.3 (3.02)
  Time spent 63-140 mg/ dL (3rd Trimester) | 68.3 (2.95) | 61.8 (3.02)
  Time spent 63-140 mg/ dL (Postpartum) | 59.0 (3.00) | 52.7 (3.02)
  Time spent >140 mg/ dL (1st Trimester) | 30.9 (3.27) | 31.9 (3.35)
  Time spent >140 mg/ dL (2nd Trimester) | 34.4 (3.27) | 40.2 (3.35)
  Time spent >140 mg/ dL (3rd Trimester) | 27.8 (3.27) | 36.4 (3.35)
  Time spent >140 mg/ dL (Postpartum) | 36.5 (3.33) | 45.7 (3.35)
  Time spent >180 mg/ dL (1st Trimester) | 12.75 (2.27) | 14.62 (2.32)
  Time spent >180 mg/ dL (2nd Trimester) | 13.05 (2.27) | 17.80 (2.32)
  Time spent >180 mg/ dL (3rd Trimester) | 8.44 (2.27) | 13.75 (2.32)
  Time spent >180 mg/ dL (Postpartum) | 15.31 (2.31) | 21.08 (2.32)

4. Primary Outcome: Fear of Hypoglycemia Score
Description: Fear of hypoglycemia is assessed as behavior, worry, and total scores of fear of hypoglycemia determined by the Hypoglycemia Fear Survey of HCL compared to SAPT in women with T1D throughout gestation and the first 4-6 weeks post-partum.
  Score Explanation: Change(s) in behavior and/or concerns of diabetics as detected by the hypoglycemia fear questionnaire. Behavior sub-scale score ranges from 10-50, with higher scores indicating more behavioral changes in the participant's daily routine to avoid low blood sugar. Worry sub-scale score ranges from 17-85, with higher scores indicating more worry or concerns because of low blood sugar. Total score ranges from 27-135, with higher scores for both sub-scales indicating more fear and a worse outcome. Subscales are added for the total scale score.
  Time Points:
  Baseline: 9 weeks gestation or earlier Visit 7: 18-20 weeks gestation Visit 10: 30-32 weeks gestation Visit 16: 4-6 weeks after delivery
Time Frame: Through study completion, an average of 9 months
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Sensor-augmented Pump Therapy (SAPT) | Hybrid Closed-loop Therapy (HCL)
Number analyzed (Participants) | 12 | 11
score on a scale
  Total Score Baseline | 69.4 (5.30) | 69.0 (5.12)
  Total Score Visit 7 | 69.0 (5.41) | 60.5 (5.27)
  Total Score Visit 10 | 67.3 (5.40) | 64.7 (5.35)
  Total Score Visit 16 (postpartum) | 68.0 (5.40) | 65.3 (5.42)
  Worry Score Baseline | 40.0 (4.26) | 39.4 (4.10)
  Worry Score Visit 7 | 38.3 (4.37) | 31.6 (4.26)
  Worry Score Visit 10 | 38.1 (4.36) | 35.9 (4.34)
  Worry Score Visit 16 (postpartum) | 38.2 (4.36) | 37.6 (4.42)
  Behavior Score Baseline | 29.8 (1.85) | 29.5 (1.79)
  Behavior Score Visit 7 | 29.9 (1.90) | 29.1 (1.89)
  Behavior Score Visit 10 | 29.0 (1.94) | 28.4 (1.89)
  Behavior Score Visit 16 (postpartum) | 29.6 (1.94) | 27.7 (2.00)

5. Secondary Outcome: Number of Episodes of Diabetic Ketoacidosis
Description: Secondary safety assessed through the number of episodes of diabetic ketoacidosis of HCL therapy compared to SAPT in women with T1D throughout gestation and the early post-partum period.
Time Frame: Through study completion, an average of 9 months
Measure: Number; unit: Number of Episodes
Arm/Group | Sensor-augmented Pump Therapy (SAPT) | Hybrid Closed-loop Therapy (HCL)
Number analyzed (Participants) | 12 | 12
Number of Episodes | 0 | 1

6. Secondary Outcome: Number of Adverse Skin Reactions
Description: Secondary safety assessed through the number of adverse skin reactions of HCL therapy compared to SAPT in women with T1D throughout gestation and the early post-partum period
Time Frame: through study completion, an average of 9 months
Measure: Number; unit: Number of Reactions
Arm/Group | Sensor-augmented Pump Therapy (SAPT) | Hybrid Closed-loop Therapy (HCL)
Number analyzed (Participants) | 12 | 12
Number of Reactions | 5 | 1

7. Secondary Outcome: Secondary Indices of Glucose Control: Mean Glucose ± Standard Deviation
Description: Secondary outcomes of indices of glycemic variability by continuous glucose monitoring as mean glucose ± standard deviation in pregnant women with T1D using HCL or SAPT therapy throughout pregnancy and early post-partum
Time Frame: through study completion, an average of 9 months
Population: The HCL group had 11 participants complete the study after randomization
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Sensor-augmented Pump Therapy (SAPT) | Hybrid Closed-loop Therapy (HCL)
Number analyzed (Participants) | 12 | 12
mg/dL
  1st Trimester | 122 (4) | 125 (4)
  2nd Trimester: number analyzed (Participants) | 12 | 11
  2nd Trimester | 126 (4) | 137 (4)
  3rd Trimester: number analyzed (Participants) | 12 | 11
  3rd Trimester | 120 (4) | 132 (4)
  Postpartum: number analyzed (Participants) | 12 | 11
  Postpartum | 130 (4) | 144 (4)

8. Secondary Outcome: Secondary Indices of Glucose Control: J-index
Description: Secondary outcomes of indices of glycemic variability by continuous glucose monitoring as J index in pregnant women with T1D using HCL or SAPT therapy throughout pregnancy and early post-partum. J index is a measure of the quality of glycemic control. Lower values represent more glycemic control and higher values represent less glycemic control.
  Formula: J-Index= 0.001 x (mean blood glucose level + SD)^2
  The J-Index has not been validated in this population of Type 1 Diabetes pregnancies.
Time Frame: through study completion, an average of 9 months
Population: The HCL group had 11 participants complete the study after randomization
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Sensor-augmented Pump Therapy (SAPT) | Hybrid Closed-loop Therapy (HCL)
Number analyzed (Participants) | 12 | 12
mg/dL
  J-Index (Run-In Phase) | 26.2 (2.25) | 29.5 (2.31)
  J-Index (1st Trimester) | 29.3 (2.25) | 32.0 (2.31)
  J-Index (2nd Trimester): number analyzed (Participants) | 12 | 11
  J-Index (2nd Trimester) | 29.5 (2.25) | 34.6 (2.31)
  J-Index (3rd Trimester): number analyzed (Participants) | 12 | 11
  J-Index (3rd Trimester) | 25.1 (2.25) | 30.7 (2.31)
  J-Index (Post-Partum): number analyzed (Participants) | 12 | 11
  J-Index (Post-Partum) | 32.1 (2.30) | 38.0 (2.31)

9. Secondary Outcome: Secondary Indices of Glucose Control: High Blood Glucose Index (HBGI)
Description: Secondary outcomes of indices of glycemic variability by continuous glucose monitoring as High Blood Glucose Index (HBGI) in pregnant women with T1D using HCL or SAPT therapy throughout pregnancy and early post-partum. HBGI is a Glucose-variability-based metric of the risk for hyperglycemia that can be calculated from CGM readings. HBGI increases with the frequency and extent of hyperglycemic excursions and has been used as a predictor of severe events. The range of values is 0-100 with 0 indicating no risk of high blood sugar and 100 indicating maximum possible risk of high blood sugar.
Time Frame: through study completion, an average of 9 months
Population: The HCL group had 11 participants complete the study after randomization
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Sensor-augmented Pump Therapy (SAPT) | Hybrid Closed-loop Therapy (HCL)
Number analyzed (Participants) | 12 | 12
score on a scale
  HBGI (Run-In Phase) | 4.54 (0.604) | 5.32 (0.618)
  HBGI (1st Trimester) | 5.23 (0.604) | 6.12 (0.618)
  HBGI (2nd Trimester): number analyzed (Participants) | 12 | 11
  HBGI (2nd Trimester) | 4.78 (0.604) | 5.61 (0.618)
  HBGI (3rd Trimester): number analyzed (Participants) | 12 | 11
  HBGI (3rd Trimester) | 3.57 (0.604) | 4.58 (0.618)
  HBGI (Post-Partum): number analyzed (Participants) | 12 | 11
  HBGI (Post-Partum) | 5.70 (0.615) | 6.42 (0.618)

10. Secondary Outcome: Secondary Indices of Glucose Control: Low Blood Glucose Index (LBGI)
Description: Secondary outcomes of indices of glycemic variability by continuous glucose monitoring as Low Blood Glucose Index (LBGI) in pregnant women with T1D using HCL or SAPT therapy throughout pregnancy and early post-partum. LBGI is a Glucose-variability-based metric of the risk for hypoglycemia. LBGI increases with the frequency and extent of hypoglycemic excursions and has been used as a predictor of severe events. The range is from 0-100 with 0 indicating no risk of low blood sugar and 100 indicating maximum possible risk of low blood sugar.
Time Frame: through study completion, an average of 9 months
Population: The HCL group had 11 participants complete the study after randomization
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Sensor-augmented Pump Therapy (SAPT) | Hybrid Closed-loop Therapy (HCL)
Number analyzed (Participants) | 12 | 12
score on a scale
  LBGI (Run-In Phase) | 5.48 (0.516) | 5.67 (0.528)
  LBGI (1st Trimester) | 5.40 (0.516) | 5.92 (0.528)
  LBGI (2nd Trimester): number analyzed (Participants) | 12 | 11
  LBGI (2nd Trimester) | 4.83 (0.516) | 4.09 (0.528)
  LBGI (3rd Trimester): number analyzed (Participants) | 12 | 11
  LBGI (3rd Trimester) | 4.06 (0.516) | 3.44 (0.528)
  LBGI (Post-Partum): number analyzed (Participants) | 12 | 11
  LBGI (Post-Partum) | 4.86 (0.525) | 3.69 (0.528)

11. Secondary Outcome: Secondary Indices of Glucose Control: Mean Amplitude of Glycemic Excursions (MAGE)
Description: Secondary outcomes of indices of glycemic variability by continuous glucose monitoring as Mean Amplitude of Glycemic Excursions (MAGE) in pregnant women with T1D using HCL or SAPT therapy throughout pregnancy and early post-partum. MAGE is the average difference between consecutive glucose peaks and nadirs greater than 1 standard deviation (SD) of the average value of glucose in a given day. Lower values represent less glycemic variability on average. Higher values represent more glycemic variability on average.
Time Frame: through study completion, an average of 9 months
Population: The HCL group had 11 participants complete the study after randomization
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Sensor-augmented Pump Therapy (SAPT) | Hybrid Closed-loop Therapy (HCL)
Number analyzed (Participants) | 12 | 12
mg/dL
  MAGE (Run-In Phase) | 84.4 (5.47) | 98.8 (5.61)
  MAGE (1st Trimester) | 91.9 (5.47) | 100.9 (5.61)
  MAGE (2nd Trimester): number analyzed (Participants) | 12 | 11
  MAGE (2nd Trimester) | 85.4 (5.47) | 94.5 (5.61)
  MAGE (3rd Trimester): number analyzed (Participants) | 12 | 11
  MAGE (3rd Trimester) | 69.2 (5.47) | 81.8 (5.61)
  MAGE (Post-Partum): number analyzed (Participants) | 12 | 11
  MAGE (Post-Partum) | 92.9 (5.59) | 99.5 (5.61)

12. Secondary Outcome: Secondary Indices of Glucose Control: Continuous Overall Net Glycemic Action (CONGAn)
Description: Secondary outcomes of indices of glycemic variability by continuous glucose monitoring as Continuous Overall Net Glycemic Action (CONGAn) in pregnant women with T1D using HCL or SAPT therapy throughout pregnancy and early post-partum. CONGAn assesses glycemic variability by calculating the difference between the glucose values taken at different timeframes. Lower values represent less glycemic differences between the timepoints. Higher values represent more glycemic differences between timepoints.
Time Frame: through study completion, an average of 9 months
Population: The HCL group had 11 participants complete the study after randomization
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Sensor-augmented Pump Therapy (SAPT) | Hybrid Closed-loop Therapy (HCL)
Number analyzed (Participants) | 12 | 12
mg/dL
  CONGAn (Run-In Phase) | 39.9 (1.99) | 42.0 (2.04)
  CONGAn (1st Trimester) | 41.3 (1.99) | 44.3 (2.04)
  CONGAn (2nd Trimester): number analyzed (Participants) | 12 | 11
  CONGAn (2nd Trimester) | 36.4 (1.99) | 40.1 (2.04)
  CONGAn (3rd Trimester): number analyzed (Participants) | 12 | 11
  CONGAn (3rd Trimester) | 29.6 (1.99) | 35.2 (2.04)
  CONGAn (Post-Partum): number analyzed (Participants) | 12 | 11
  CONGAn (Post-Partum) | 40.0 (2.03) | 42.6 (2.04)

13. Secondary Outcome: Medical Outcomes Study (MOS) Short-Form 36 Score
Description: Quality of life as measured by scores from the MOS Short-Form 36 (quality of life) of HCL and SAPT arms in pregnant women with T1D. The SF-36 has eight scaled scores; the scores are weighted sums of the questions in each section. Scores range from 0 - 100 Lower scores = more disability, higher scores = less disability Sections: Vitality, Physical functioning, Bodily pain, General health perceptions, Physical role functioning, Emotional role functioning, Social role functioning, Mental health
Time Frame: through study completion, an average of 9 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Sensor-augmented Pump Therapy (SAPT) | Hybrid Closed-loop Therapy (HCL)
Number analyzed (Participants) | 12 | 12
score on a scale
  SF36 Total (1st Trimester) | 73.96 (3.51) | 82.23 (3.44)
  SF36 Total (2nd Trimester) | 76.30 (3.80) | 85.72 (4.04)
  SF36 Total (3rd Trimester) | 66.01 (3.92) | 77.09 (4.04)
  SF36 Total (Postpartum) | 70.45 (4.09) | 80.55 (4.05)
  SF36 General Health (1st Trimester) | 63.33 (4.40) | 64.05 (4.32)
  SF36 General Health (2nd Trimester) | 62.61 (4.60) | 67.77 (4.69)
  SF36 General Health (3rd Trimester) | 59.95 (4.67) | 62.72 (4.69)
  SF36 General Health (Postpartum) | 64.70 (4.77) | 65.45 (4.69)
  SF36 Pain (1st Trimester) | 81.33 (4.68) | 90.66 (4.62)
  SF36 Pain (2nd Trimester) | 85.94 (5.32) | 93.89 (5.74)
  SF36 Pain (3rd Trimester) | 63.37 (5.52) | 80.78 (5.75)
  SF36 Pain (Postpartum) | 67.50 (5.80) | 79.64 (5.75)
  SF36 Social Functioning (1st Trimester) | 85.99 (3.89) | 90.36 (3.86)
  SF36 Social Functioning (2nd Trimester) | 81.62 (4.54) | 95.31 (4.96)
  SF36 Social Functioning (3rd Trimester) | 82.28 (4.74) | 89.83 (4.96)
  SF36 Social Functioning (Postpartum) | 82.14 (5.00) | 91.26 (4.97)
  SF36 Emotional Wellbeing (1st Trimester) | 78.59 (3.61) | 83.18 (3.56)
  SF36 Emotional Wellbeing (2nd Trimester) | 70.45 (4.07) | 84.15 (4.37)
  SF36 Emotional Wellbeing (3rd Trimester) | 76.12 (4.22) | 78.72 (4.38)
  SF36 Emotional Wellbeing (Postpartum) | 71.42 (4.42) | 84.56 (4.38)
  SF36 Energy (1st Trimester) | 46.22 (5.48) | 53.06 (5.39)
  SF36 Energy (2nd Trimester) | 51.04 (5.99) | 57.29 (6.32)
  SF36 Energy (3rd Trimester) | 48.56 (6.16) | 45.97 (6.32)
  SF36 Energy (Postpartum) | 40.95 (6.40) | 53.76 (6.33)
  SF36 Emotional Limits (1st Trimester) | 81.98 (7.33) | 95.74 (7.20)
  SF36 Emotional Limits (2nd Trimester) | 84.70 (8.01) | 98.44 (8.55)
  SF36 Emotional Limits (3rd Trimester) | 76.96 (8.28) | 91.08 (8.56)
  SF36 Emotional Limits (Postpartum) | 84.51 (8.65) | 98.00 (8.57)
  SF36 Physical Health Limits (1st Trimester) | 71.70 (8.96) | 88.61 (8.82)
  SF36 Physical Health Limits (2nd Trimester) | 83.72 (10.16) | 95.69 (10.97)
  SF36 Physical Health Limits (3rd Trimester) | 42.62 (10.45) | 90.26 (10.98)
  SF36 Physical Health Limits (Postpartum) | 81.83 (10.99) | 81.83 (10.99)
  SF36 Physical Functioning (1st Trimester) | 88.89 (4.22) | 93.47 (4.18)
  SF36 Physical Functioning (2nd Trimester) | 91.52 (4.86) | 93.31 (5.28)
  SF36 Physical Functioning (3rd Trimester) | 79.65 (5.06) | 78.97 (5.28)
  SF36 Physical Functioning (Postpartum) | 84.69 (5.32) | 92.15 (5.29)

14. Secondary Outcome: INSPIRE Questionnaire Score
Description: Quality of life as measured by scores from the INSPIRE questionnaire of HCL in pregnant women with T1D. The INsulin Dosing Systems: Perceptions, Ideas, Reflections, and Expectations (INSPIRE) is a survey consisting of 22 questions that assess user expectations and experiences with automated insulin delivery systems. Scores are calculated by determining the mean of the sum of all questions then multiplying the mean by 25 for a range of 0 to 100. Higher scores indicate more positive perceptions of the system. Each survey question uses a 5 point Likert scale ranging from 0 (strongly disagree) to 4 (strongly agree).
Time Frame: through study completion, an average of 9 months
Population: INSPIRE Questionnaire only among HCL randomized group
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Hybrid Closed-loop Therapy (HCL)
Number analyzed (Participants) | 12
score on a scale
  Baseline/1st Trimester | 73.6 (4.1)
  2nd Trimester | 79.3 (4.8)
  3rd Trimester | 76.2 (4.6)
  Post-Partum | 76.5 (4.8)

15. Secondary Outcome: Insulin Delivery Satisfaction Survey (IDSS) Score
Description: Device acceptability as measured by scores from the Insulin Delivery Satisfaction Survey of HCL and SAPT arms in pregnant women with T1D. The IDSS scale has a total score and 3 subscales: effective, burdensome, and inconvenient. Possible scores range from 1-5, with higher scores indicating higher satisfaction with insulin delivery system. Scores are reflective of the mean of the Total or subscale questions.
Time Frame: through study completion, an average of 9 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Sensor-augmented Pump Therapy (SAPT) | Hybrid Closed-loop Therapy (HCL)
Number analyzed (Participants) | 12 | 12
score on a scale
  IDSS Total (1st Trimester) | 4.00 (0.14) | 4.06 (0.14)
  IDSS Total (2nd Trimester) | 3.80 (.015) | 4.19 (0.16)
  IDSS Total (3rd Trimester) | 3.85 (0.16) | 3.92 (0.16)
  IDSS Total (Postpartum) | 3.92 (0.16) | 4.20 (0.16)
  IDSS Effective (1st Trimester) | 4.12 (0.15) | 4.16 (0.15)
  IDSS Effective (2nd Trimester) | 4.13 (0.17) | 4.32 (0.18)
  IDSS Effective (3rd Trimester) | 4.26 (0.17) | 4.16 (0.18)
  IDSS Effective (Postpartum) | 4.26 (0.18) | 4.32 (0.18)
  IDSS Burdensome (1st Trimester) | 2.10 (0.19) | 2.08 (0.19)
  IDSS Burdensome (2nd Trimester) | 2.46 (0.21) | 2.04 (0.22)
  IDSS Burdensome (3rd Trimester) | 2.36 (0.21) | 2.24 (0.22)
  IDSS Burdensome (Postpartum) | 2.41 (0.22) | 2.06 (0.22)
  IDSS Inconvenient (1st Trimester) | 2.03 (0.18) | 1.90 (0.18)
  IDSS Inconvenient (2nd Trimester) | 2.27 (0.20) | 1.69 (0.21)
  IDSS Inconvenient (3rd Trimester) | 2.36 (0.21) | 2.17 (0.21)
  IDSS Inconvenient (Postpartum) | 2.07 (0.22) | 1.63 (0.21)

16. Secondary Outcome: Glucose Monitoring Satisfaction Survey (GMSS) Score
Description: Device acceptability as measured by scores from the Glucose Monitoring Satisfaction Survey questionnaires of HCL compared to SAPT in pregnancy women with T1D. The GMSS has a total score and 4 subscales: openness, emotional burden, behavioral burden, and trust. Possible scores range from 1-5, with higher total scores indicating greater satisfaction. Scores are reflective of the mean of the Total or subscale questions.
Time Frame: through study completion, an average of 9 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Sensor-augmented Pump Therapy (SAPT) | Hybrid Closed-loop Therapy (HCL)
Number analyzed (Participants) | 12 | 12
score on a scale
  GMSS Total (1st Trimester) | 4.07 (0.13) | 3.83 (0.13)
  GMSS Total (2nd Trimester) | 3.65 (0.15) | 4.06 (0.16)
  GMSS Total (3rd Trimester) | 3.66 (0.15) | 3.89 (0.16)
  GMSS Total (Postpartum) | 3.90 (0.16) | 3.95 (0.16)
  GMSS Trust (1st Trimester) | 3.99 (0.19) | 3.65 (0.20)
  GMSS Trust (2nd Trimester) | 3.43 (0.22) | 4.10 (0.24)
  GMSS Trust (3rd Trimester) | 3.75 (0.23) | 4.10 (0.24)
  GMSS Trust (Postpartum) | 3.76 (0.24) | 3.77 (0.24)
  GMSS Behavioral Burden (1st Trimester) | 1.86 (0.15) | 2.01 (0.15)
  GMSS Behavioral Burden (2nd Trimester) | 2.07 (0.17) | 1.78 (0.18)
  GMSS Behavioral Burden (3rd Trimester) | 2.29 (0.17) | 1.99 (0.18)
  GMSS Behavioral Burden (Postpartum) | 1.99 (0.18) | 1.97 (0.18)
  GMSS Emotional Burden (1st Trimester) | 1.83 (0.19) | 2.11 (0.19)
  GMSS Emotional Burden (2nd Trimester) | 2.41 (0.21) | 1.85 (0.22)
  GMSS Emotional Burden (3rd Trimester) | 2.34 (0.22) | 1.92 (0.22)
  GMSS Emotional Burden (Postpartum) | 2.06 (0.23) | 2.02 (0.23)
  GMSS Openness (1st Trimester) | 3.95 (0.14) | 3.74 (0.14)
  GMSS Openness (2nd Trimester) | 3.58 (0.16) | 3.76 (0.18)
  GMSS Openness (3rd Trimester) | 3.55 (0.17) | 3.43 (0.18)
  GMSS Openness (Postpartum) | 3.86 (0.18) | 3.97 (0.18)

17. Secondary Outcome: Maternal Outcomes: Number of Participants With Preeclampsia/Eclampsia
Description: Maternal outcomes includes preeclampsia/eclampsia in pregnant women with T1D using HCL therapy compared to those using SAPT throughout gestation and in the early post-partum period
Time Frame: through study completion, an average of 9 months
Measure: Count of Participants; unit: Participants
Arm/Group | Sensor-augmented Pump Therapy (SAPT) | Hybrid Closed-loop Therapy (HCL)
Number analyzed (Participants) | 12 | 11
Participants | 4 | 4

18. Secondary Outcome: Maternal Outcomes: Number of Participants With Cesarean Delivery
Description: Maternal outcomes includes cesarean delivery in pregnant women with T1D using HCL therapy compared to those using SAPT throughout gestation and in the early post-partum period
Time Frame: through study completion, an average of 9 months
Measure: Count of Participants; unit: Participants
Arm/Group | Sensor-augmented Pump Therapy (SAPT) | Hybrid Closed-loop Therapy (HCL)
Number analyzed (Participants) | 12 | 11
Participants | 10 | 7

19. Secondary Outcome: Maternal Outcomes: Average Gestational Weight Gain
Description: Maternal outcomes includes gestational weight gain in pregnant women with T1D using HCL therapy compared to those using SAPT throughout gestation and in the early post-partum period
Time Frame: through study completion, an average of 9 months
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Sensor-augmented Pump Therapy (SAPT) | Hybrid Closed-loop Therapy (HCL)
Number analyzed (Participants) | 12 | 11
kg | 14.1 (6.0) | 11.5 (4.1)

20. Secondary Outcome: Fetal Outcomes: Number of Participants With a Fetal Loss (Miscarriage or Stillbirth)
Description: Fetal outcomes includes fetal loss (miscarriage or stillbirth) in pregnant women with T1D using HCL therapy compared to those using SAPT throughout gestation and in the early post-partum period
Time Frame: through study completion, an average of 9 months
Measure: Count of Participants; unit: Participants
Arm/Group | Sensor-augmented Pump Therapy (SAPT) | Hybrid Closed-loop Therapy (HCL)
Number analyzed (Participants) | 12 | 11
Participants | 0 | 0

21. Secondary Outcome: Fetal Outcomes: Number of Infants With Large-for-gestational Age Outcome
Description: Fetal outcomes includes large-for-gestational age in pregnant women with T1D using HCL therapy compared to those using SAPT throughout gestation and in the early post-partum period
Time Frame: through study completion, an average of 9 months
Measure: Count of Participants; unit: Participants
Arm/Group | Sensor-augmented Pump Therapy (SAPT) | Hybrid Closed-loop Therapy (HCL)
Number analyzed (Participants) | 12 | 11
Participants | 6 | 6

22. Secondary Outcome: Fetal Outcomes: Number of Participants With Neonatal Hypoglycemia Infants
Description: Fetal outcomes includes neonatal hypoglycemia in pregnant women with T1D using HCL therapy compared to those using SAPT throughout gestation and in the early post-partum period
Time Frame: through study completion, an average of 9 months
Measure: Count of Participants; unit: Participants
Arm/Group | Sensor-augmented Pump Therapy (SAPT) | Hybrid Closed-loop Therapy (HCL)
Number analyzed (Participants) | 12 | 11
Participants | 4 | 5

ADVERSE EVENTS:
Time Frame: through study completion, an average of 9 months
Arm/Group | Sensor-augmented Pump Therapy (SAPT) | Hybrid Closed-loop Therapy (HCL)
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12 | 6/12
Other Adverse Events (participants affected / at risk) | 10/12 | 11/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sensor-augmented Pump Therapy (SAPT) (N=12) | Hybrid Closed-loop Therapy (HCL) (N=12)
Fetal Demise (Pregnancy, puerperium and perinatal conditions) | 0 | 1 (1) — Fetal demise one day after randomization into the HCL group
DKA (Endocrine disorders) | 0 | 1 (1) — Diabetic Ketoacidosis
Severe Hypoglycemia (Endocrine disorders) | 0 | 1 (1)
Preeclampsia with Severe Features (Cardiac disorders) | 0 | 2 (2)
Chronic Hypertension with Superimpose Preeclampsia with Severe Features (Cardiac disorders) | 0 | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Sensor-augmented Pump Therapy (SAPT) (N=12) | Hybrid Closed-loop Therapy (HCL) (N=12)
Miscarriage (Pregnancy, puerperium and perinatal conditions) | 2 | 0 — Pre-viable pregnancy loss
Polyhydramnios (Pregnancy, puerperium and perinatal conditions) | 2 (3) | 2 (2)
Preterm Birth (Pregnancy, puerperium and perinatal conditions) | 2 (2) | 2 (2) — Delivery before 37 weeks gestation
Hyperglycemia (Endocrine disorders) | 1 (1) | 3 (4)
Ketonuria (Endocrine disorders) | 3 (3) | 1 (1)
Hypoglycemia (Endocrine disorders) | 0 | 2
Gestational Hypertension (Cardiac disorders) | 3 | 1
Preeclampsia without Severe Features (Cardiac disorders) | 1 | 1
Illness (Infections and infestations) | 5 | 2 — Cold, COVID-19 infection, Upper Respiratory Illness/Infection, Respiratory Virus, Sinus Infection
Sensor Site Irritation (Product Issues) | 5 | 1 — Bleeding, Bruising or Skin Irritation at Sensor Site
Post-Partum Depression/Anxiety (Psychiatric disorders) | 0 | 1/11 — The HCL group had 11 participants complete the study after randomization due to a fetal loss in one participant 1 day after randomization.
Anemia (Blood and lymphatic system disorders) | 1 | 0
Hypothyroidism (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Musculoskeletal or Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Headache/Migraine (General disorders) | 1 (1) | 3 (4)
Ovarian Cyst (Reproductive system and breast disorders) | 1 | 0
Nausea/Vomiting (Pregnancy, puerperium and perinatal conditions) | 0 | 4
Gastroesophageal Reflux Disease (Gastrointestinal disorders) | 1 | 1
Large for Gestational Age Infant (General disorders) | 2 | 1/11 — The HCL group had 11 participants complete the study after randomization due to a fetal loss in one participant 1 day after randomization.
Yeast Infection (Reproductive system and breast disorders) | 0 | 1 (2)
Tenosynovitis (General disorders) | 1 | 0
Mastitis (Reproductive system and breast disorders) | 1 (2) | 1 (1)
Neonatal Hypoglycemia (General disorders) | 0 | 1/11 — The HCL group had 11 participants complete the study after randomization due to a fetal loss in one participant 1 day after randomization.
Seasonal Allergies (Immune system disorders) | 1 (2) | 0
Vaginal Aching (Reproductive system and breast disorders) | 0 | 1
Infant Respiratory Distress (General disorders) | 2 | 2/11 — The HCL group had 11 participants complete the study after randomization due to a fetal loss in one participant 1 day after randomization.
Abdominal Pain (General disorders) | 2 | 0
Post-Partum Pain (Pregnancy, puerperium and perinatal conditions) | 0 | 1/11 — The HCL group had 11 participants complete the study after randomization due to a fetal loss in one participant 1 day after randomization.
Pelvic Pain (General disorders) | 0 | 1
Mild Post-Partum Hypertension (Cardiac disorders) | 1 | 0
Food Poisoning (Gastrointestinal disorders) | 0 | 1
Cholestasis (Hepatobiliary disorders) | 0 | 1
Ankle/Feet Swelling (General disorders) | 1 | 2
Carpal Tunnel (Nervous system disorders) | 1 | 0
Foot Pain (General disorders) | 1 | 0
Placental Hemorrhage (Pregnancy, puerperium and perinatal conditions) | 0 | 1
Fetal Arrhythmia (Cardiac disorders) | 1 | 0
Fetal Bradycardia (Cardiac disorders) | 1 | 0
Blood Ketones (Endocrine disorders) | 1 | 0
Increased Fetal Movement (Pregnancy, puerperium and perinatal conditions) | 1 | 0
Infant Gastroesophageal Reflux Disease (Gastrointestinal disorders) | 1 | 0
Infant Laryngomalacia/ Supraglottic Edema (General disorders) | 1 | 0
Short Cervix (Reproductive system and breast disorders) | 1 | 0
Hip Soreness (Musculoskeletal and connective tissue disorders) | 1 | 0
Leg Bruising (General disorders) | 1 | 0 — Not related to sensor site placement
Vaginal Bleeding (Reproductive system and breast disorders) | 0 | 1
Elevated Blood Pressure (Mild) (Cardiac disorders) | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1
Infant Shoulder Dystocia (General disorders) | 0 | 1
Hives (Immune system disorders) | 0 | 1
Finger Wart (General disorders) | 0 | 1
Abnormal Ultrasound Findings (General disorders) | 0 | 1
Scratched Cornea (Eye disorders) | 0 | 1
Eczema Flare-Up (Skin and subcutaneous tissue disorders) | 0 | 1
Non-Reassuring Fetal Wellbeing (General disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-01-19): https://cdn.clinicaltrials.gov/large-docs/86/NCT03774186/Prot_SAP_000.pdf